CLINICAL TRIAL: NCT02609867
Title: A Feasibility Study to Evaluate the Safety and Effectiveness of Implantation of 'Flowise Cerebral Flow Diverter' for the Treatment of Unruptured Wide-necked Cerebral Aneurysm in the Internal Carotid Artery
Brief Title: A Feasibility Study to Evaluate the Safety and Effectiveness of Implantation of Flowise Cerebral Flow Diverter (Flowise)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDV-001
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flowise Cerebral Flow Diverter (Experimental): Flowise Cerebral Flow Diverter (TaeWoong Medical Co., Ltd. Korea)
  Interventions: Device: Flowise Cerebral Flow Diverter

INTERVENTIONS:
Device: Flowise Cerebral Flow Diverter — Flowise Cerebral Flow Diverter Placement

SUMMARY:
The purpose of this study is to evaluate the safety and short-term effectiveness of implantation of 'Flowise Cerebral Flow Diverter' for the treatment of unruptured wide-necked cerebral aneurysm in the internal carotid artery.

DETAILED DESCRIPTION:
Flowise is indicated for use in patients with unruptured wide-necked aneurysm in the internal carotid artery. Consecutive subject data should be collected at discharge, 1, 3, and 6 month post Flowise implantation.

ELIGIBILITY:
Inclusion Criteria:

* Functional neurological state ≤2 mRS
* Unruptured wide-neck aneurysm in the internal carotid artery has a size >8mm, a neck ≥4mm, or dome/neck ratio <2
* Parent artery with diameter ≥3.25mm and ≤4.5mm
* Patient willing to provide written informed consent and comply with follow-up requirements

Exclusion Criteria:

* Intracranial hemorrhage within 30 days
* Untreated ruptured intracranial aneurysm
* ≥1 intracranial aneurysm except the target one requires treatment within 6 months
* Immunosuppressive disease
* Active infectious disease (e.g. endocarditis, meningitis)
* Platelet count < 100 x 103 cells/mm3
* Female of child-bearing potential who are unable to take adequate contraceptive precautions, are known to be pregnant, or are currently breastfeeding an infant.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-22 (Actual)

PRIMARY OUTCOMES:
Procedural success | 5days
  Procedural success is defined as the full expansion of the Flowise identified on angiography and the full coverage of the targeted aneurysm neck in the absence of periprocedural stroke or death.
≥50% intracranial aneurysm size reduction success at 6 month | 6months
  Intracranial aneurysm size is measured by Transfemoral Cerebral Angiography (TFCA).
Aneurysm occlusion success at 6month | 6months
  Aneurysm occlusion success is defined as Raymond class Ⅰ, Ⅱ

SECONDARY OUTCOMES:
≥50% Parent artery stenosis or occlusion | 6months
Newly developed neurological disorder | 6months
  Newly developed neurological disorder is defined as neurological problem lasts for at least 1 month post procedure and ≥3 modified Rankin Scale (mRS).
Ipsilateral stroke | 6months
  Ipsilateral stroke is defined as ≥5 according to the National Institute of Health Stroke Scale (NIHSS).
30-day death | 6months
  30-day death was defined as death within 30 days post procedure.
Other adverse events | 6months

CONTACTS AND LOCATIONS:
Overall Officials: Buyng Moon Kim, PhD. MD, Principal Investigator — Yonsei University Healthcare System, Severance Hospital
Locations (1):
- Yonsei University Healthcare System, Severance Hospital, Seoul, Yeonsei-ro Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided